CLINICAL TRIAL: NCT06569030
Title: Effect of Spinal Orthosis on Sagittal and Frontal Parameters in Adolescent Idiopathic Scoliosis
Brief Title: Effect Spinal Orthosis on Sagittal and Frontal Parameters in Scoliosis
Acronym: SpinalOrthosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yılmaz, Research Assistant (Orthotist and Prosthetist), Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: mervearslann
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; Scoliosis Brace; 3D spine analysis; plantar pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with Adolescent Idiopathic Scoliosis Who Receive Spinal Orthosis (Other)
  Interventions: Biological: spinal orthoses

INTERVENTIONS:
Biological: spinal orthoses — Evaluation of scoliosis treatment in people using spinal orthoses

SUMMARY:
It has been observed that there are insufficient studies on whether the conservative treatment of AIS with Chêneau spinal orthosis provides 3D correction on the scoliotic curve and its effect on the spine and lower extremity parameters. The aim of this study is to investigate the effect of Chêneau spinal orthosis application on sagittal and frontal parameters at 3 and 6 months follow-up in adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a three-dimensional deformity of the spine that is commonly seen in individuals aged 10-18 years, and spinal orthosis application, one of the conservative treatment methods, is widely preferred today. Lyon, Milwaukee, Gensingen, Boston and Rigo System Chêneau spinal orthoses are among the most frequently preferred today. Rigo system Chêneau (RCS) spinal orthosis aims to correct scoliosis in 3D in sagittal, transverse and coronal planes. Studies have indicated that spinal orthosis application may have limited corrective effect on sagittal and transverse planes scoliotic curvature. In order to obtain the most effective result in spinal orthosis application, it is important to fully understand the connection mechanisms between different planes and their relationship with the lower extremity. It has been observed that studies on whether conservative treatment of spinal orthosis in adolescent idiopathic scoliosis (AIS) can provide 3D correction on the scoliotic curve and its effect on spine and lower extremity parameters are insufficient. AIS individuals who will undergo Chêneau type spinal orthosis application that meets the inclusion criteria will be included in the study. Demographic information of the participants will be obtained with a patient information form and a scoliosis assessment form. Radiographs are planned to be obtained using an EOS (EOS-imaging®, Paris, France) imaging device, which is a low-dose imaging device that provides simultaneous anterior-posterior and lateral views while standing. Spine and lower extremity parameters will be evaluated from the obtained images. Plantar pressure and balance assessment is planned to be performed with a DIERS Pedoscan device connected to the DIERS Formetric system. SRS-22 (Scoliosis Research Society-22) questionnaire is planned to be used in the assessment of the quality of life of the individuals. Brace Questionnaire is planned to be used in the assessment of spinal orthosis satisfaction. All data will be evaluated by statistical analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 years old
* Cobb angle: 15-45°
* Individuals with AIS who will be using a Chêneau type spinal orthosis for the first time • Spinal orthosis recommended for at least 18 hours per day
* Risser ≤ 3

Exclusion Criteria:

* Using a foot orthosis
* Neurological problem
* Surgery history
* Lower extremity length difference greater than 1 cm

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
EOS-imaging® | Change from Baseline of treatment at 3 and 6 months
  Radiographs were planned to be obtained using an EOS (EOS-imaging®, Paris, France) imaging device, which is a low-dose imaging device that provides simultaneous anterior-posterior and lateral views in the standing position. Spine and lower extremity parameters will be evaluated from the obtained image.
  Spine parameters; cervical lordosis ( C1C3, C2C6, C3C7), pelvic oblique, pelvic coronal obliquity angle, thoracolumbar kyphosis, lumbar lordosis, pelvic incidence, pelvic tilt, sacral slope, sagittal vertical angle, coronal vertical angle will be evaluated.
  Lower Extremity Parameters; hip-knee-ankle angle, medial proximal femoral angle, mechanical lateral distal femoral angle, medial proximal tibial angle, lateral distal tibial angle, lower extremity length, femur length, tibia length, recurvation angle of the knee joint will be measured.
Spine Rotation Measurement | Change from Baseline of treatment at 3 and 6 months
  Trunk Rotation Measurement: Scoliometer; is used during the person's "Adam's Forward Bend Test" to determine the trunk rotation angle.
DIERS Formetric Pedoscan | Change from Baseline of treatment at 3 and 6 months
  Plantar Pressure and Balance Assessment It is planned to be performed with the DIERS Pedoscan device connected to the DIERS Formetric system in plantar pressure and balance assessment. DIERS Pedoscan allows the assessment of foot pressure distribution while standing. It is preferred for measuring plantar pressure changes during the individual's bipedal static stance and walking. There are static, dynamic, postural balance analysis methods in pedobarographic assessment. Numerical data is obtained for foot analysis with these methods.
Scoliosis Research Society (SRS-22 test) | Change from Baseline of treatment at 3 and 6 months
  assessment of quality of life SRS-22 is a scale used to assess the quality of life in individuals with spinal deformity.
Brace Questionnaire (BrQ) | Change from Baseline of treatment at 3 and 6 months
  Evaluation of Spinal Orthosis Satisfaction Brace Questionnaire (BrQ) is a questionnaire used to measure the effect of brace treatment on quality of life in adolescent idiopathic scoliosis.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yılmaz, Study Director — https://www.medipol.edu.tr/
Locations (1):
- Acıbadem Üniversitesi Maslak Hastanesi Omurga Sağlık Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No